CLINICAL TRIAL: NCT01369147
Title: Comparative Effectiveness of Energy Doses in Critical Illness
Brief Title: The Energy Dose Study
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was halted pending additional funding and ultimately was terminated due to difficulties with ongoing recruitment, etc.
Sponsor: Emory University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Thomas R. Ziegler, Professor of Medicine, Emory University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: IRB00049495; 1R21DK089369 (NIH)
Record Dates: First submitted 2011-05-25; First posted 2011-06-08 (Estimated); Results first posted 2022-06-10 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-05

CONDITIONS: Critical Illness
Keywords: Surgical Intensive Care Unit (SICU); Calories; Total Parenteral Nutrition (TPN); Tube Feeding; Optimum Energy Dose in SICU; Malnutrition; Hospital-acquired Infection
MeSH Terms: conditions — Critical Illness; Hyperphagia; Malnutrition; Cross Infection | interventions — Parenteral Nutrition; Propofol; clevidipine; Enteral Nutrition

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Parenteral nutrition energy dose at 0.6 x measured REE (Experimental): Participants in this study arm will be provided a total daily calorie (kcal) intake at 0.6 x REE for up to 28 days. The dose of parenteral nutrition (PN) will be adjusted taking into account any calories from propofol, clevidipine, dextrose-containing IV fluids surpassing 500 mL/day, and any enteral feedings, to obtain the energy dose that the participant was randomized to receive.
  Interventions: Drug: Parenteral Nutrition; Drug: Propofol; Drug: Clevidipine; Drug: Dextrose-containing IV Fluids; Drug: Enteral feeding
- Parenteral nutrition energy dose at 1.0 x measured REE (Active Comparator): Participants in this study arm will be provided a total daily calorie (kcal) intake at 1.0 x REE for up to 28 days. The dose of PN will be adjusted taking into account any calories from propofol, clevidipine, dextrose-containing IV fluids surpassing 500 mL/day, and any enteral feedings, to obtain the energy dose that the participant was randomized to receive.
  Interventions: Drug: Parenteral Nutrition; Drug: Propofol; Drug: Clevidipine; Drug: Dextrose-containing IV Fluids; Drug: Enteral feeding
- Parenteral nutrition energy dose at 1.3 x measured REE (Experimental): Participants in this study arm will be provided a total daily calorie (kcal) intake at 1.3 x REE for up to 28 days. The dose of PN will be adjusted taking into account any calories from propofol, clevidipine, dextrose-containing IV fluids surpassing 500 mL/day, and any enteral feedings, to obtain the energy dose that the participant was randomized to receive.
  Interventions: Drug: Parenteral Nutrition; Drug: Propofol; Drug: Clevidipine; Drug: Dextrose-containing IV Fluids; Drug: Enteral feeding

INTERVENTIONS:
Drug: Parenteral Nutrition — The PN dose will be written for each 24-hr period taking into account any kilocalories (kcal) provided as part of standard of care from propofol, clevidipine, dextrose-containing IV fluid exceeding 500 mL/day, and enteral feedings.
Drug: Propofol — The PN dose will be written for each 24-hr period taking into account calories provided as lipid emulsion in the sedative propofol (1.1 kcal/mL).
  Other Names: Diprivan
Drug: Clevidipine — The PN dose will be written for each 24-hr period taking into account calories provided as lipid emulsion in clevidipine (2 kcal/mL).
  Other Names: Cleviprex
Drug: Dextrose-containing IV Fluids — The PN dose will be written for each 24-hr period taking into account calories provided from dextrose-containing IV fluid orders exceeding 500 mL/day.
Drug: Enteral feeding — Enteral nutrition is caloric intake through the gastrointestinal (GI) tract via food consumed through the mouth or a feeding tube delivering nutrition directly to the stomach or small intestines. The PN dose will be written for each 24-hr period taking into account calories provided from any enteral feedings.

SUMMARY:
The investigators have designed this single-center Randomized Clinical Trial (RCT) to prospectively compare, for the first time, the clinical efficacy of different energy doses in intensive care unit (ICU) patients requiring parenteral nutrition (PN) due to intestinal failure/dysfunction. This study intends to enroll a total of 60 patients (20 per energy dose group) to generate critical preliminary data needed to inform subsequent appropriately powered Phase III multicenter trials.

DETAILED DESCRIPTION:
Protein and/or energy deficits are associated with increased rates of hospital infection, skeletal muscle weakness, impaired wound healing, and prolonged convalescence in ICU patients. To prevent or treat malnutrition, enteral nutrition (EN) and/or parenteral nutrition (PN) are routinely given worldwide to a significant proportion of ICU patients. Optimal caloric requirements in critically ill patients are unknown due to a lack of rigorous randomized clinical trials. The comparative efficacy of energy doses in critically ill patients is unknown and clinical recommendations are conflicting and controversial.

The primary aim of this study is to perform a controlled, double-blind, prospective, randomized, intent-to-treat Phase II clinical trial to test the efficacy of three specific energy doses on 28-day total hospital-acquired infections (primary endpoint), blood stream infections (BSI), and other important clinical outcomes in medical/surgical ICU patients requiring specialized parenteral ± enteral feeding. The investigators would also determine the impact of cumulative and mean daily 28-day energy deficits on clinical outcome endpoints; the practical utility of estimated resting energy expenditure (REE) determined by Harris-Benedict equation versus measured REE across different energy doses. The investigators would also like to determine the impact of administered energy dose and energy deficits on global metabolomic patterns over time and their association with key clinical outcomes.

Participants will be randomized to receive one of three specific energy doses, 0.6, 1.0 and 1.3 times measured REE, given for 28 consecutive days during the ICU and post-ICU course.

ELIGIBILITY:
Inclusion Criteria:

* A signed informed consent is in place on the patient's chart
* The patient is at least 18 but not more than 90 years of age at time of ICU admission
* The patient has a body mass index (BMI) less than 40 kg/m^2
* The patient has been admitted to either a medical or surgical (non-neurological) ICU and is expected to survive and remain in the ICU for at least 72 hours after entry
* There is central venous access for administration of the study PN
* The patient's primary physician(s) will allow the investigative team to manage the study PN and enteral feedings during the current hospitalization
* The patient is expected to require total or partial central venous PN for 7 or more subsequent days after entry on a clinical basis

Exclusion Criteria:

* The patient is pregnant
* The patient has unresuscitated clinical sepsis, defined as unstable blood pressure despite vasopressor support and mean arterial pressure (MAP) < 60 mm Hg on at least 3 consecutive readings within a 3-hour period during the 24 hours prior to study entry
* The patient was admitted to the ICU following trauma or burns
* The patient has significant renal dysfunction (defined as serum creatinine > 2.5 mg/dL or deemed to have significant acute kidney injury by the primary physicians) and is not receiving continuous renal replacement therapy (CRRT) or intermittent hemodialysis
* The patient has previously undergone an organ transplantation
* The patient has a current malignancy or is currently receiving an active regimen of chemotherapy and/or radiotherapy to treat a previously diagnosed malignancy
* The patient has a history of HIV/AIDS
* The patient has received any investigational drug within 60 days prior to study entry
* The patient is unable or unwilling to participate in study procedures such as longitudinal blood draws and administration of study nutrient formulations

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-07 (Actual); Primary Completion 2014-12-02 (Actual); Study Completion 2014-12-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R Ziegler, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Parenteral Nutrition Energy Dose at 0.6 x Measured REE: Participants in this study arm were provided a total daily calorie (kcal) intake at 0.6 x resting energy expenditure (REE) for up to 28 days. The dose of parenteral nutrition (PN) was adjusted taking into account any calories from propofol, clevidipine, dextrose-containing IV fluids surpassing 500 mL/day, and any enteral feedings, to obtain the energy dose that the participant was randomized to receive.
- Parenteral Nutrition Energy Dose at 1.0 x Measured REE: Participants in this study arm were provided a total daily calorie (kcal) intake at 1.0 x REE for up to 28 days. The dose of parenteral nutrition (PN) was adjusted taking into account any calories from propofol, clevidipine, dextrose-containing IV fluids surpassing 500 mL/day, and any enteral feedings, to obtain the energy dose that the participant was randomized to receive.
- Parenteral Nutrition Energy Dose at 1.3 x Measured REE: Participants in this study arm were provided a total daily calorie (kcal) intake at 1.3 x REE for up to 28 days. The dose of parenteral nutrition (PN) was adjusted taking into account any calories from propofol, clevidipine, dextrose-containing IV fluids surpassing 500 mL/day, and any enteral feedings, to obtain the energy dose that the participant was randomized to receive.
Period: Overall Study
Arm/Group | Parenteral Nutrition Energy Dose at 0.6 x Measured REE | Parenteral Nutrition Energy Dose at 1.0 x Measured REE | Parenteral Nutrition Energy Dose at 1.3 x Measured REE
Started | 3 | 5 | 4
Completed | 3 | 4 | 4
Not Completed | 0 | 1 | 0
Not completed — All collected data were unintentionally destroyed | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: This analysis includes participants who have baseline data available; all data were unintentionally destroyed for one participant assigned to the 1.0 REE group.
Groups:
- Parenteral Nutrition Energy Dose at 0.6 x Measured REE: Participants in this study arm were provided a total daily calorie (kcal) intake at 0.6 x REE for up to 28 days. The dose of parenteral nutrition (PN) was adjusted taking into account any calories from propofol, clevidipine, dextrose-containing IV fluids surpassing 500 mL/day, and any enteral feedings, to obtain the energy dose that the participant was randomized to receive.
- Total: Total of all reporting groups
Arm/Group | Parenteral Nutrition Energy Dose at 0.6 x Measured REE | Parenteral Nutrition Energy Dose at 1.0 x Measured REE | Parenteral Nutrition Energy Dose at 1.3 x Measured REE | Total
Number analyzed (Participants) | 3 | 4 | 4 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.05 (21.50) | 60.56 (14.90) | 51.73 (11.20) | 53.66 (15.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3 | 6
  Male | 2 | 2 | 1 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 4 | 4 | 11
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 2 | 3
  White | 2 | 4 | 2 | 8
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 4 | 4 | 11
Acute Physiologic Assessment and Chronic Health Evaluation II (APACHE II) Score [Count of Participants; unit: Participants] — The APACHE II score is an assessment of hospital mortality risk based on 14 physiological characteristics including patient age, prior health history, and current physiological measurements. Total scores range from 0 to 71 where higher scores indicate increasing risk of hospital death. Scores below 15 are associated with a mortality rate of less than 25%, while scores of 15 and above are associated with a mortality rate of greater than 25% that increases as the APACHE II score increases. Scores of 35 and above are associated with a hospital mortality rate of 85%.
  Participants
    APACHE II Score of 15 or Less | 1 | 2 | 2 | 5
    APACHE II Score Greater Than 15 | 2 | 2 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Hospital-acquired Infection
Description: The number of participants with a hospital-acquired infection during the study period is presented here.
Time Frame: Up to Day 28
Population: This analysis includes participants with complete data available.
Measure: Count of Participants; unit: Participants
Arm/Group | Parenteral Nutrition Energy Dose at 0.6 x Measured REE | Parenteral Nutrition Energy Dose at 1.0 x Measured REE | Parenteral Nutrition Energy Dose at 1.3 x Measured REE
Number analyzed (Participants) | 3 | 4 | 4
Participants | 1 | 0 | 1

2. Secondary Outcome: Number of Participants With Bloodstream Infection
Description: The count of participants acquiring a bloodstream infection during the study period is presented here.
Time Frame: Up to Day 28
Population: This analysis includes participants with complete data available.
Measure: Count of Participants; unit: Participants
Arm/Group | Parenteral Nutrition Energy Dose at 0.6 x Measured REE | Parenteral Nutrition Energy Dose at 1.0 x Measured REE | Parenteral Nutrition Energy Dose at 1.3 x Measured REE
Number analyzed (Participants) | 3 | 4 | 4
Participants | 1 | 0 | 0

3. Secondary Outcome: Ventilator Free Days
Description: The mean number of ICU ventilator-free days among participants.
Time Frame: Up to Day 28
Population: This analysis includes participants with complete data available.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Parenteral Nutrition Energy Dose at 0.6 x Measured REE | Parenteral Nutrition Energy Dose at 1.0 x Measured REE | Parenteral Nutrition Energy Dose at 1.3 x Measured REE
Number analyzed (Participants) | 3 | 4 | 4
days | 20.67 (9.45) | 19.75 (3.40) | 17.25 (9.32)

4. Secondary Outcome: Number of Days in Intensive Care Unit (ICU)
Description: The ICU length of stay (in days) is presented here for each study arm.
Time Frame: Up to 28 Days
Population: This analysis includes participants with complete data available.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Parenteral Nutrition Energy Dose at 0.6 x Measured REE | Parenteral Nutrition Energy Dose at 1.0 x Measured REE | Parenteral Nutrition Energy Dose at 1.3 x Measured REE
Number analyzed (Participants) | 3 | 4 | 4
days | 7.33 (3.21) | 14.25 (14.75) | 4.00 (1.41)

5. Secondary Outcome: Number of Days in Hospital
Description: The hospitalization length of stay (in days) is presented here for each study arm.
Time Frame: Up to Day 28
Population: This analysis includes participants with complete data available.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Parenteral Nutrition Energy Dose at 0.6 x Measured REE | Parenteral Nutrition Energy Dose at 1.0 x Measured REE | Parenteral Nutrition Energy Dose at 1.3 x Measured REE
Number analyzed (Participants) | 3 | 4 | 4
days | 27.33 (1.15) | 25.00 (3.56) | 17.75 (9.25)

6. Other Pre Specified Outcome: Cumulative 28-day Energy Deficit
Description: The daily energy deficit of kilocalories was calculated by subtracting the calculated mean daily Measured Resting Energy Expenditure (measured using a metabolic cart) from the actual daily energy intake obtained from participant nutrition intake records. The cumulative energy deficit is the sum of daily energy deficits during the time participants were hospitalized, up to 28 days.
Time Frame: Up to Day 28
Population: This analysis includes participants with complete data available.
Measure: Mean (Standard Deviation); unit: kilocalories (kcal)
Arm/Group | Parenteral Nutrition Energy Dose at 0.6 x Measured REE | Parenteral Nutrition Energy Dose at 1.0 x Measured REE | Parenteral Nutrition Energy Dose at 1.3 x Measured REE
Number analyzed (Participants) | 3 | 4 | 4
kilocalories (kcal) | 2631 (3076.04) | 11511.50 (14765.43) | 2414.75 (1562.65)

7. Other Pre Specified Outcome: Mean Daily Energy Deficit
Description: The daily energy deficit of kilocalories was calculated by subtracting the calculated mean daily Measured Resting Energy Expenditure (measured using a metabolic cart) from the actual daily energy intake obtained from participant nutrition intake records. The mean daily energy deficit was calculated during the time participants were hospitalized, up to 28 days.
Time Frame: Up to Day 28
Population: This analysis includes participants with complete data available.
Measure: Mean (Standard Deviation); unit: kcal/day
Arm/Group | Parenteral Nutrition Energy Dose at 0.6 x Measured REE | Parenteral Nutrition Energy Dose at 1.0 x Measured REE | Parenteral Nutrition Energy Dose at 1.3 x Measured REE
Number analyzed (Participants) | 3 | 4 | 4
kcal/day | 647.33 (561.46) | 1065.75 (716.01) | 1076.50 (613.34)

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected from the time of participant entry into the study through the end of study participation, up to 28 days.
Description: Collection of non-serious adverse events was limited to those that were expected among ICU patients receiving parenteral nutrition and tube feeding, specifically: clinically significant pulmonary aspiration, pneumothorax, development of worsening renal function with serum creatinine > 5.0 mg/dL or requiring new initiation of renal replacement therapy, development of severe hepatic dysfunction (serum total serum bilirubin > 15.0 mg/dL), hyperglycemia > 250 mg/dL, and hypoglycemia < 50 mg/dL.
Arm/Group | Parenteral Nutrition Energy Dose at 0.6 x Measured REE | Parenteral Nutrition Energy Dose at 1.0 x Measured REE | Parenteral Nutrition Energy Dose at 1.3 x Measured REE
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/3 | 0/4 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-06-02): https://cdn.clinicaltrials.gov/large-docs/47/NCT01369147/Prot_SAP_000.pdf